CLINICAL TRIAL: NCT02099916
Title: Prospective Randomized Trial on the Effect of DHEA Administration in Women With Poor Ovarian Reserve Undergoing Controlled Ovarian Stimulation for IVF. Impact on Stimulation Characteristics and and Pregnancy Outcome.
Brief Title: Administration of DHEA in Patients With Poor Response to Ovarian Stimulation for IVF
Acronym: DHEA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Athens (Other)
Collaborators: Lito Maternity Hospital (Other)
Responsible Party: Principal Investigator, Nikos Vlahos, Associate Professor of Obstetrics and Gynecology, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NV04222014
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Efficacy of DHEA; Pregnancy Rate; Diminished Ovarian Reserve; Changes in AMH
Keywords: DHEA, pregnancy, ovarian reserve, AMH
MeSH Terms: interventions — Gonadotropins; Dehydroepiandrosterone; Menotropins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gonadotropins plus DHEA (Active Comparator): Patients in this group will be stimulated according to a short stimulation protocol with gonadotropins and GnRH antagonists. Prior to the stimulation will be treated with DHEA 25 mg PO tid for 12 weeks.
  Interventions: Drug: gonadotropins plus DHEA; Drug: Gonadotropins
- Gonadotropins (Active Comparator): Patients in this group will be stimulated according to a short stimulation protocol with gonadotropins and GnRH antagonists.
  Interventions: Drug: gonadotropins plus DHEA; Drug: Gonadotropins

INTERVENTIONS:
Drug: gonadotropins plus DHEA — Women in the DHEA group will received 25 mg of DHEA three times a day for at least 12 weeks.
  Other Names: DHEA
Drug: Gonadotropins — All patients will be stimulated with a fixed GnRH-antagonist protocol. Ovarian stimulation will be initiated with 450 IU of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH.
  Other Names: Menopur 75IU, Gonal

SUMMARY:
Poor responders to ovarian stimulation represents one of the most frustrating problems in reproductive medicine. The investigators hypothesize that ovarian response of those patients could improve by treating these patients with 25 mg DHEA tid for 12 weeks prior to stimulation.

DETAILED DESCRIPTION:
Patients diagnosed with poor ovarian response will be included in the study. The definition of poor response was based on the presence of at least one of the following criteria: Age > 40 years old, day 2 FSH >9.5 mIU/ml, AMH < 2ng/ml ,at least one previous COH with less than 3 oocytes retrieved, at least one cancelled attempt due to poor response, estradiol less than 500 pg/ml on the day of HCG. All patients will be counseled regarding their prognosis and other treatment options including oocyte donation as well as adoption were also presented and discussed in detail. All patients will be aware that the use of DHEA is experimental and informed consent was obtained for those agreeing to use the medication. Women in the DHEA group will receive 25 mg of DHEA three times a day for at least 12 weeks. During this period, women will be subjected to monthly measurements of early follicular phase FSH and estradiol. Anti-Mullerian Hormone (AMH) will be measured prior to the initiation of treatment and at the end of the observation period. Patients will be stimulated with a short GnRH-antagonist protocol. Briefly, all women will have measurements of serum FSH and estradiol and a pelvic sonogram on the second day of their cycle. Providing that serum FSH is < 17 mIU/ml and estradiol is < 70 pg/ml on day 2 , ovarian stimulation will be initiated with 450 IU of gonadotropins either in the form of a combination of highly purified urinary FSH and LH or with a combination of Rec FSH and Rec LH. All patients will be re-evaluated on day 5 of the stimulation, and dosage adjustments will be made and the antagonists (Cetrorelix or ganirelix 0.25 mg/day) will be initiated. When at least 2 follicles reach an average diameter of 17 mm, final oocyte maturation will be triggered with 10,000IU of hCG ( Pregnyl, Organon, Greece Inc.). Oocyte retrieval will be performed 34 to 36 hours later. All patients will undergo ICSI. Patients with successful fertilization will have embryo transfer under sonographic guidance on day 3 after retrieval.

ELIGIBILITY:
Inclusion Criteria:

* Women with poor response to ovarian stimulation. The definition of poor response was based on the presence of at least one of the following criteria: Age > 40 years old, day 2 FSH >9.5 mIU/ml, AMH < 2ng/ml ,at least one previous COH with less than 3 oocytes retrieved, at least one cancelled attempt due to poor response, estradiol less than 500 pg/ml on the day of HCG.

Exclusion Criteria:

* All other women that do not fulfill the above mentioned criteria

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | At 12 weeks after DHEA administration and at 18 months
  At the completion of the ovarian stimulation patients that will proceed to transfer and have a positive pregnancy test will have sonographic evaluation for confirmation of clinical pregnancy.

SECONDARY OUTCOMES:
changes in ovarian reserve indexes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Vlahos, AssProfessor, Study Chair — University of Athens, 2nd Department of Obstetrics and Gynecology